CLINICAL TRIAL: NCT03890250
Title: Investigation of the Effectiveness of Neuromuscular Electrical Stimulation in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Neuromuscular Electrical Stimulation in Patients With Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other); Istanbul University (Other)
Responsible Party: Principal Investigator, Buket AKINCI, Assistant Proffesor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018/12-1
Record Dates: First submitted 2019-03-13; First posted 2019-03-26 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Idiopathic Pulmonary Fibrosis; Neuromuscular Electrical Stimulation
Keywords: pulmonary rehabilitation; neuromuscular electrical stimulation
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Thirty IPF patients aged 40-80 years who are followed up at Istanbul University, Istanbul Medical Faculty Chest Disease Department will include in the study. Participants will be divided into two groups as the NMES group and the Sham Training Group, using a computer-assisted randomization table.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The assessor will be blind to the randomization and the investigator will be blind to the results of assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham group (Sham Comparator): Following the assessments, sham group will participate in a 20-30 minute low-medium intensity aerobic exercise training with cycling ergometer. In Sham training group, NMES will be applied to the same region after aerobic exercise, current frequency is 5 Hz, current transit time is 300 μs, 10 seconds warning, 30 seconds electrical stimulation in 20 seconds rest period. The rehabilitation program will be administered two days a week for 8 weeks under the supervision of a physiotherapist.
  Interventions: Other: Aerobic exercise
- NMES group (Experimental): Following the assessments, both groups will participate in a 20-30 minute low-medium intensity aerobic exercise training with cycling ergometer.
  After the aerobic exercise in NMES group, bilateral NMES application on Quadriceps femoris muscle will be applied as symmetrical biphasic square wave current with a wave frequency of 35-60 Hz, phase transition time of 8 seconds and active resting time of 15 seconds.
  Interventions: Other: Aerobic exercise; Other: Neuromuscular electrical stimulation

INTERVENTIONS:
Other: Aerobic exercise — A 20-30 minutes low-medium intensity aerobic exercise training with cycling ergometer.
Other: Neuromuscular electrical stimulation — Bilateral NMES application on Quadriceps femoris muscle will be applied as symmetrical biphasic square wave current with a wave frequency of 35-60 Hz, phase transition time of 8 seconds and active resting time of 15 seconds
  Arms: NMES group

SUMMARY:
Pulmonary rehabilitation should be initiated and lifelong at the time of diagnosis for patients with IPF. However, the symptoms of the disease and its progression limit clinical options in terms of participation and sustainability in rehabilitation programs. For this purpose, patients with IPF need physiotherapy and rehabilitation options that will not increase the symptoms associated with exercise and contribute to the program in the long term. Neuromuscular electrical stimulation (NMES) is a rehabilitation option that can be applied to specific muscle groups without the ventilator and cardiac load especially in patients who can not actively exercise or have decreased muscle strength. In adult patients with an advanced disease characterized by reduced muscle strength, the use of NMES in addition to aerobic exercise programs is recommended as part of rehabilitation programs. In the literature, no studies investigating the efficacy of NMES have been found in individuals with IPF or interstitial lung disease. NMES application in addition to aerobic exercise seems to be a reasonable option when considering the symptoms of patients with IPF and the progression of the disease. The aim of this project is to investigate the efficacy of NMES in addition to aerobic exercise in IPF patients based on evidence by objective methods.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) is a progressive, fibrotic interstitial lung disease characterized by progressive dyspnoea, reduced exercise capacity, quality of life, and classified as a rare disease. With the increase in medical treatment options, the progression of the disease slows down. Increased time of survival has increased the need for pulmonary rehabilitation programs that have been shown to be effective in patients' exercise capacity, participation in daily living activities, and improvement in the quality of life. Patients with IPF have been shown to be able to improve dyspnoea, fatigue, exercise capacity, daily living activities and quality of life with home-based or supervised breathing, posture, strengthening and aerobic/endurance exercise programs.

Pulmonary rehabilitation should be initiated and lifelong at the time of diagnosis for patients with IPF. However, the symptoms of the disease and its progression limit clinical options in terms of participation and sustainability in rehabilitation programs. For this purpose, patients with IPF need physiotherapy and rehabilitation options that will not increase the symptoms associated with exercise and contribute to the program in the long term. Neuromuscular electrical stimulation (NMES) is a rehabilitation option that can be applied to specific muscle groups without the ventilator and cardiac load especially in patients who can not actively exercise or have decreased muscle strength. In adult patients with an advanced disease characterized by reduced muscle strength, the use of NMES in addition to aerobic exercise programs is recommended as part of rehabilitation programs. In the literature, no studies investigating the efficacy of NMES have been found in individuals with IPF or interstitial lung disease. NMES application in addition to aerobic exercise seems to be a reasonable option when considering the symptoms of patients with IPF and the progression of the disease. The aim of this project is to investigate the efficacy of NMES in addition to aerobic exercise in IPF patients based on evidence by objective methods.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of IPF according to current ATS / ERS guidelines has been followed by a pulmonary specialist for at least 6 months
* Patients who are clinically stable, have no flare or infection.

Exclusion Criteria:

* Orthopedic and neurological problems that may interfere with exercise training,
* Modification of medical treatment during the study,
* Unstable cardiac diseases,
* Participation in another pulmonary rehabilitation program over the past 12 months,
* Inadequate cooperation,
* Contraindications for the application of neuromuscular electrical stimulation (risk of embolism, neoplasm, infection in the region of application, pacemaker, sensory defect).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Assessment of exercise capacity | 2 months
  Exercise capacity will be assessed with 6-minutes walk test. The six minutes walking distance will be recorded in "metres".
Assessment of endurance capacity | 2 months
  Endurance capacity will be assessed with "Shuttle Endurance Walking test". The number of shuttles will be recorded and maximum VO2 will be calculated.

SECONDARY OUTCOMES:
Assessment of peripheral muscle strength | 2 months
  Peripheral muscle strength will be assessed with hand held dynamometer for quadriceps muscles.
Assessment of fatigue | 2 months
  Fatigue will be assessed with Fatigue Severity Scale. The scale consists 9 questions. The minimum score is 0 and maximum score is 63. Higher scores indicate worse fatigue level.
Assessment of activities of daily living | 2 months
  The activities of daily living will be assessed by "The London Chest Daily Activities of Daily Living Questionnaire. The scale has 4 subgroups; self-care (4 question), about home (six question), physical activity (2 question) and leisure time (3 question). The minimum score is 0 and maximum score is 75. Higher scores indicate worse conditions.
Assessment of quality of life: "Saint George Quality of Life Survey | 2 months
  The quality of life will be assessed by "Saint George Quality of Life Survey". The scale consists 50 questions. The minimum score is 0 and the maksimum score is 100. Higher scores indicate poor quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Buket Akıncı, Assist.Prof., Principal Investigator — Biruni University
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Holland AE, Wadell K, Spruit MA. How to adapt the pulmonary rehabilitation programme to patients with chronic respiratory disease other than COPD. Eur Respir Rev. 2013 Dec;22(130):577-86. doi: 10.1183/09059180.00005613. PMID 24293474
- [Result] Jones S, Man WD, Gao W, Higginson IJ, Wilcock A, Maddocks M. Neuromuscular electrical stimulation for muscle weakness in adults with advanced disease. Cochrane Database Syst Rev. 2016 Oct 17;10(10):CD009419. doi: 10.1002/14651858.CD009419.pub3. PMID 27748503